CLINICAL TRIAL: NCT01915056
Title: A Pilot Study of a Geriatric Assessment Intervention for Older Cancer Patients Receiving Chemotherapy
Brief Title: A Geriatric Assessment Intervention for Older Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Supriya Mohile, Supriya Gupta Mohile, M.D., M.S. - Associate Professor of Medicine at the James Wilmot Cancer Center at the University of Rochester. Director, Geriatric Oncology Clinic., University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCCO-13034
Record Dates: First submitted 2013-07-23; First posted 2013-08-02 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Cancer
Keywords: Comprehensive Geriatric Assessment (CGA); GA-driven interventions; Toxicity; Outcomes; providing information; older cancer patients; first-line chemotherapy; second-line chemotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (No Intervention): Control Arm = Standard of Care. Patients who are randomized to the control arm will only have abnormal results on Geriatric Depression Scale (GDS) and cognitive evaluation communicated to their primary oncologist, as is customary. These results will be communicated to the primary team via electronic medical record and/or email communication. No other summary will be provided to oncologist.
- Treatment Arm (Experimental): Treatment Arm = Standard care plus GA results and recommendations. For patients assigned to the treatment arm, individuals will be offered the option of completing the GA during a visit with their primary oncologist, or attending an additional visit at the multidisciplinary geriatric oncology clinic (GA-driven intervention). The intervention consists of providing results of geriatric assessment in a summary to oncologists.
  Interventions: Other: GA-driven Intervention

INTERVENTIONS:
Other: GA-driven Intervention — For patients assigned to the treatment arm, individuals will be offered the option of completing the GA during a visit with their primary oncologist, or attending an additional visit at the multidisciplinary geriatric oncology clinic. The intervention consists of providing results of geriatric assessment in a summary to oncologists.
  Arms: Treatment Arm

SUMMARY:
The purpose of this study is to determine whether information regarding GA and GA-driven interventions improves outcomes in older cancer patients receiving first-line or second-line chemotherapy by comparing rates of chemotherapy toxicity, hospitalizations, dose delays and early termination of treatment in patients with and without GA-driven interventions. The investigators will identify information that will be useful based on questionnaire responses and blood tests. These results will be used to better understand which recommendations and interventions will benefit older cancer patients. It is our hope that these tools, which are well-established at identifying areas of risk, will provide meaningful opportunities for intervention to promote your safety during cancer management. The investigators will be able to use this information to teach others on how to best care for adults aged 70 and older with cancer.

DETAILED DESCRIPTION:
Although cancer is very common in older patients, the optimal treatment for cancer for this subset of patients is not well established. As a result of lack of knowledge on the safety and efficacy of chemotherapy in older adults, a significant proportion of older patients receiving chemotherapy have toxicity. There is also little information regarding how to best make decisions for and implement interventions to improve outcomes of older patients with cancer who are to receive treatment. Additionally, there is marked heterogeneity in the geriatric population, and patients of similar chronologic age may have wide disparity in their overall health status. Geriatricians utilize a tool called the Geriatric Assessment (GA) to gauge an older patient's overall health status and identify potential areas of deficits. The GA is a comprehensive tool, incorporating the assessment of physical function, co-morbid conditions, social support, nutritional, psychological, and cognitive status and medication review. A small number of studies in the oncology literature have demonstrated the value of GA in guiding cancer-directed treatment plans for older patients. GA can identify potential areas of deficits in an older patient's overall health status that have been shown to predict chemotherapy toxicity and guide interventions to improve outcomes for older patients. Studies of interventions in community-dwelling older adults have demonstrated efficacy at improving deficits identified on GA. However, in older patients with cancer, there is currently limited data regarding how GA can affect decision-making for treatment and impact overall clinical care.

In a two-arm, randomized pilot study, we will evaluate the effect of GA and GA-driven interventions on the outcomes of older cancer patients receiving first-line or second-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of solid tumor malignancy or lymphoma
* Have advanced cancer
* Have received a recommendation for first or second line treatment with chemotherapy by their primary oncologist. Treatment regimens may include chemotherapy, chemoradiotherapy, targeted agents or monoclonal antibody.
* Planned chemotherapy for at least 3 months
* Be age 70 or older
* Have a live expectancy with treatment of 6 months or greater
* Able to provide informed consent or, if the physician deems the patient to not have decision-making capacity, a patient-designated health care proxy (that was pre-existing; prior to the patient losing decision-making capacity) must sign consent per institutional (University of Rochester and Research Subject Review Board) policies on consent for incapacitated/decisionally impaired subjects164,165
* Able to read and understand English (or possess a designated health care proxy that can do the same that was designated prior to the patient losing decision-making capabilities)

Exclusion Criteria:

* Have surgery planned within 3 months of consent
* Have a planned referral to the geriatric oncology clinic within one month of treatment initiation
* Patients who do not have decision-making capacity (decisionally or cognitively impaired) AND do NOT have a previously designated health care proxy (established prior to their cognitive impairment) available to sign consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Chemotherapy Toxicity | Over 3 months
  The primary outcome measure for this study is to determine if GA-driven interventions improve outcomes in older cancer patients receiving first-line or second-line chemotherapy by comparing rates of chemotherapy toxicity, hospitalizations, dose delays and early termination of treatment. The primary analysis will be a comparison of the proportion of patients who developed grade >3 toxicity over 3 months time using the likelihood ratio test.

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Mohile, MD, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - Highland Hospital, Rochester, New York
  - Pluta Cancer Center, Rochester, New York
  - University of Rochester Wilmot Cancer Center, Rochester, New York